CLINICAL TRIAL: NCT00088192
Title: An Open Label, Non-Comparative Protocol for Use of Intravitreous Pegaptanib Sodium Injection Every 6 Weeks in Patients With Exudative Age-Related Macular Degeneration (AMD)
Brief Title: Intravitreous Pegaptanib Sodium Injection in Patients With Exudative Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eyetech Pharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EOP1010
Record Dates: First submitted 2004-07-21; First posted 2004-07-22 (Estimated); Last update posted 2005-08-30 (Estimated); Status verified 2005-08

CONDITIONS: Macular Degeneration
Keywords: AMD; Age-Related Macular Degeneration; Exudative Subfoveal Age Related Macular Degeneration with Subfoveal Choroidal Neovascularization
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

INTERVENTIONS:
Drug: pegaptanib sodium

SUMMARY:
To provide Pegaptanib sodium injection to patients with subfoveal choroidal neovascularization (CNV) secondary to AMD, who are unable to participate in any of the Sponsor's other clinical studies with this drug for AMD, until such time as the patient's lesion is considered to have resolved or stabilized in the opinion of the treating ophthalmologist, or product becomes commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity in the study eye between 20/40 and 20/320.
* Subfoveal choroidal neovascularization, secondary to age related macular degeneration, with a total lesion size [including blood, scar/atrophy & neovascularization] of < 12 total disc areas, of which at least 50% must be active CNV.
* Any subretinal hemorrhage must comprise no more than 50% of total lesion size.

General Criteria:

* Patients of either gender, aged greater than 50 years.
* Women must be using two forms of effective contraception, or be post-menopausal for at least 12 months prior to study entry, or surgically sterile. If of child-bearing potential, a serum pregnancy test must be performed within 48 hours prior to treatment and the result made available prior to treatment initiation. The two forms of effective contraception must be implemented during the study and for at least 60 days following the last dose of test medication.
* Written informed consent.

Exclusion Criteria:

* Any subfoveal scarring or atrophy and no more than 25% of the total lesion size may be made up of scarring or atrophy.
* Patients who are eligible for PDT with Visudyne
* Patients who are eligible for any other of the Sponsor's ongoing AMD studies still open to enrollment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-07

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Doheny Eye Institute, Los Angeles, California
  - Connecticut Retina Consultants, L.L.C., Bridgeport, Connecticut
  - New England Retina Associates, Hamden, Connecticut
  - Retina Health Center, Fort Myers, Florida
  - Retina Associates, New Orleans, Louisiana
  - Cumberland Valley Retina Center, Hagerstown, Maryland
  - New England Eye Center, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Associated Retinal Consultants, Royal Oak, Michigan
  - Eye Foundation of Kansas City, Kansas City, Missouri
  - The Eye Center of Concord, Concord, New Hampshire
  - Vitreo- Retinal Assoc. of NJ, Belleville, New Jersey
  - Retina Associates of New Jersey, P.A., Teaneck, New Jersey
  - L.I. Vitreo-Retinal Consultants, Great Neck, New York
  - Retina Associates of Cleveland Inc., Lakewood, Ohio
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - The Casey Eye Institute, Portland, Oregon
  - Palmetto Retina Center, Columbia, South Carolina
  - Valley Retina Associates, P.A., McAllen, Texas
  - University of Vermont College of Medicine, Burlington, Vermont

REFERENCES:
- See also: Sponsors Website — http://www.eyetech.com